CLINICAL TRIAL: NCT04087096
Title: Denosumab to Prevent High-Turnover Bone Loss After Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of California, San Francisco (Other); San Francisco VA Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elaine W. Yu, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20187525; 20187525 (Other Grant/Funding Number: Amgen - Investigator Sponsored Study)
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Bariatric Surgery Candidate; Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Denosumab (Experimental): Denosumab 60mg subcutaneous injection every 6 months
  Interventions: Drug: Denosumab; Drug: Zoledronic Acid
- Placebo (Placebo Comparator): Placebo subcutaneous injection every 6 months
  Interventions: Drug: Placebo; Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Denosumab — Denosumab will be administered at postoperative months 1, 7, and 13
  Other Names: Prolia
  Arms: Denosumab
Drug: Placebo — Placebo will be administered at postoperative months 1, 7, and 13
  Arms: Placebo
Drug: Zoledronic Acid — Zoledronic Acid 5mg will be administered intravenously at postoperative month 19
  Other Names: Reclast

SUMMARY:
Bariatric surgery leads to bone loss and increases fracture risk. This study evaluates whether denosumab can prevent the high-turnover bone loss that occurs after Roux-en-Y Gastric Bypass (RYGB) and sleeve gastrectomy (SG) surgery.

DETAILED DESCRIPTION:
Bariatric surgery is a highly effective weight loss treatment, but one of the unintended side effects of these procedures is high-turnover bone loss and metabolic bone disease. Denosumab is a monoclonal antibody to RANKL that acts as a potent inhibitor of bone resorption. The investigators are conducting a randomized placebo-controlled trial to evaluate the ability of denosumab to prevent bone loss after RYGB or SG surgery in older adults. At the conclusion of the study, all participants will be given zoledronic acid.

ELIGIBILITY:
Inclusion criteria:

* Postmenopausal women who are planning RYGB or SG surgery
* Men aged ≥ 50 years who are planning RYGB or SG surgery

Exclusion criteria:

* Prior bariatric surgery
* Weight = 400 lbs (due to limitations of bone imaging equipment)
* Renal disease
* Hypercalcemia or hypocalcemia
* Hypomagnesemia
* Serum 25-OH vitamin D (25OHD) < 20 ng/mL
* Hyperparathyroidism
* Liver disease (AST or ALT > 2 x upper normal limit)
* HCT < 32%
* History of malignancy (except basal cell carcinoma) in the past 1 year
* Significant cardiopulmonary disease
* Major psychiatric disease
* History of celiac disease or inflammatory bowel disease
* Excessive alcohol or substance abuse
* Paget's disease, primary hyperparathyroidism, or any other known congenital or acquired bone disease other than osteoporosis
* Current hyperthyroidism or use of levothyroxine with TSH < 0.1 uIU/mL
* Current use of loop diuretics
* Current use or use in the past 12 months of oral bisphosphonates or DMAB
* Current use or use within the past 3 months of SERMs or calcitonin
* Current use or use within the past 3 months of estrogen
* Use of testosterone therapy if dose has changed within the last 3 months, or if dose change or discontinuation is planned in the upcoming 18 months
* Any current or previous use of teriparatide, strontium, or any parenteral bisphosphonate
* Use of oral or parenteral glucocorticoids for more than 14 days within the past 6 months
* Extensive dental work involving extraction or dental implant within the past 2 months or planned in the upcoming 18 months
* DXA BMD T-score of < -3.0 at PA spine, total hip, or femoral neck
* Current use of anti-VEGF drug

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tabira T. [Immunological abnormalities in multiple sclerosis]. No To Shinkei. 1983 Jun;35(6):535-41. No abstract available. Japanese. PMID 6194805
- [Background] Ramirez-Lassepas M, Quinones MR. Heparin therapy for stroke: hemorrhagic complications and risk factors for intracerebral hemorrhage. Neurology. 1984 Jan;34(1):114-7. doi: 10.1212/wnl.34.1.114. PMID 6537834
- [Background] Marina Fiol C. [Treatment of the hepatic repercussions of cholelithiasis]. Minerva Med. 1966 Jul 14;57(56):2550-2. No abstract available. Italian. PMID 6002877

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Denosumab | Placebo
Started | 24 | 12
Completed | 24 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab | Placebo | Total
Number analyzed (Participants) | 24 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.71 (5.03) | 56.58 (10.04) | 56.67 (6.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 9 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 22 | 10 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 17 | 11 | 28
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 12 | 36
Pre-Op Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 43.9 (5.59) | 43.8 (6.36) | 43.87 (5.76)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Total Hip Bone Mineral Density
Time Frame: Pre-operative baseline to post-operative month 19
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Denosumab | Placebo
Number analyzed (Participants) | 24 | 12
percentage of change | 0.60 [-0.66 to 1.87] | -6.44 [-8.74 to -4.13]

ADVERSE EVENTS:
Time Frame: Baseline to 19 months
Arm/Group | Denosumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/12
Serious Adverse Events (participants affected / at risk) | 5/24 | 1/12
Other Adverse Events (participants affected / at risk) | 24/24 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab (N=24) | Placebo (N=12)
Musculoskeletal Issues (Musculoskeletal and connective tissue disorders) | 2 | 0
Vaccine Reaction (General disorders) | 1 | 0
Orthostasis (General disorders) | 0 | 1
Other GI Issues (Gastrointestinal disorders) | 2 | 0
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab (N=24) | Placebo (N=12)
Musculoskeletal Issues (Musculoskeletal and connective tissue disorders) | 22 | 11
Skin Rash or Discomfort (Skin and subcutaneous tissue disorders) | 12 | 4
Tingling/numbness (Nervous system disorders) | 9 | 5
Nausea (Gastrointestinal disorders) | 2 | 0
Other GI Issues (Gastrointestinal disorders) | 6 | 2
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 2
Dental Issues (General disorders) | 6 | 4
COVID infection (Infections and infestations) | 5 | 3
Confusion (General disorders) | 3 | 1
Lightheadedness/dizziness (General disorders) | 5 | 1
Abnormal Labs (Investigations) | 3 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Depression (Psychiatric disorders) | 2 | 0
Eye Irritation (Eye disorders) | 1 | 1
Eye Procedure (Surgical and medical procedures) | 2 | 0
Headache (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT04087096/Prot_SAP_000.pdf